CLINICAL TRIAL: NCT05608239
Title: Prospective, Single-site, Open Label Study to Assess the Safety and Efficacy of Injectable Poly-L-Lactic Acid (Sculptra Aesthetic) for Volume Loss in the Temples Using Dual Plane Injections
Brief Title: Safety and Efficacy of Injectable Poly-L-Lactic Acid for Volume Loss in the Temples Using Dual Plane Injections
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sadick Research Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SadickRG
Record Dates: First submitted 2022-11-02; First posted 2022-11-08 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Lipoatrophy; Aging
MeSH Terms: conditions — Lipodystrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sculptra® Aesthetic (Experimental)
  Interventions: Device: Sculptra aesthetic

INTERVENTIONS:
Device: Sculptra aesthetic — The goal of the study is to evaluate the volumizing and bio-stimulatory effects of sculptra injections in the temples with total volume of the diluted product as 9 ml (8 ml of sterile water and 1 ml of Lidocaine).

SUMMARY:
Temporal volume loss is part of the natural aging process of the face. It is primarily the consequence of fat pad atrophy, but bone loss, ligament weakening, soft tissue, and muscle also contribute. . The goal of the study is to evaluate the volumizing and bio-stimulatory effects of sculptra injections in the temples.

DETAILED DESCRIPTION:
This is a prospective, single-site, open label study to assess the safety and efficacy of injectable Poly-L-Lactic Acid (Sculptra aesthetic) for volume loss in the temples using dual plane injections. Eligible subjects will get up to 3 treatments four weeks apart with poly-L-lactic acid, (Sculptra) in the temples. After the treatments, subjects will return to the research site 1 month and 6 months post last treatment for follow up visits.Eligible subjects will get up to 3 treatment sessions 4 weeks apart with ether Sculptra® Aesthetic or saline following a randomized list. During the study period, subjects will return to the research site for visits at 5 and 6 months post baseline (±7 days).

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are able to give voluntary, written informed consent to participate in this study and from whom consent has been obtained including HIPAA authorization
* Healthy males or females over 25 years old with temporal hollows volume deficit of Grade 2 to 4 on the Galderma Temple Volume Deficit Scale
* Subjects with Fitzpatrick photo skin types I-IV
* Subjects who agree not to have any procedures affecting facial wrinkles (e.g. filler, botulinum toxin, radiofrequency, laser, intense-pulsed light, ultrasound) for the duration of the study
* Subjects who do agree not to have any other procedures affecting skin quality (microdermabrasion, peels, acne treatments, etc.) for the duration of the study
* Subjects who understand this study and are able to follow study instructions and are willing to attend the required study visits
* Subjects who agree to be photographed for research reasons and their identity may not be concealed in these photographs.

Exclusion Criteria:

* Subjects who are pregnant, planning to become pregnant or breastfeeding. A urine pregnancy test will be done to rule out pregnancy
* Subjects of child-bearing potential who are not using an approved method of birth control (oral contraceptives, intrauterine device, contraceptive implant, barrier methods with spermicide or abstinence). Females of non-childbearing potential are defined as post-menopausal (absence of menstrual bleeding for one year), hysterectomy or bilateral oophorectomy.
* Subjects who cannot understand or are not willing to comply with the requirements of the study
* Subjects who have a known allergy to poly-L-lactic acid, carboxymethylcellulose, non-pyrogenic mannitol or any anesthetic
* Subjects who have taken any NSAIDs (aspirin, ibuprofen, etc.) within 7 days before treatment
* Subjects who have taken acetaminophen 24 hours before treatment
* Subjects who have had fillers or botulinum toxin in the treatment area in the past 12 months
* Subjects who have had treatments with poly-L-lactic acid in the face at any time
* Subjects who have had any kind of facial dermabrasion, chemical peel, laser, or IPL treatment including superficial treatments for aesthetic reasons in the past 6 months or for the duration of the study
* Subjects who does not agree to avoid using tanning beds or intensive exposure to the sun 2 two weeks prior to each office visit.
* Subjects who have any dermatologic conditions including acne, rosacea, eczema, psoriasis, actinic keratosis, severe sun damage, infection or scars within the treatment area
* Subjects who have an active inflammatory process (skin eruptions such as cysts, pimples, rashes or hives) or infection within the treatment area
* Subjects who have any known cancer including skin cancers (basal cell carcinoma, squamous cell carcinoma and melanoma)
* Subjects who have had systemic corticosteroid therapy in the past 6 months or for the duration of the study
* Subjects with a known history of poor wound healing
* Subjects with a known history of keloids (excessive scarring)
* Subjects who are HIV positive
* Subjects who have an existing medical condition that the Investigator considers may put the subject at risk or compromise their participation in the study
* Subjects who have participated in another research study in the past 30 days
* Subjects who are currently involved in any injury litigation claims

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-11 (Estimated); Primary Completion 2023-07 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Clinical evaluation of PLLA injection for efficacy, to restore the volume loss in temporal area | 16 weeks
  at least one degree of improvement in the temporal area volume using the Galderma Temple Volume Deficit Scale (Moradi et al Dermatol Surg. 2020 Sep;46(9): 1148-1154) and GAIS at the last follow up as compared to baseline.

SECONDARY OUTCOMES:
Improvement of facial skin laxity | 16 weeks
  Improvement of facial skin laxity will be defined as at least 1 point of improvement in the facial area using the 10-point facial laxity rating scale (Silva Hector, Dermatol Surg.2016 Dec;42(12):1370-1379) from baseline throughout week 36.
Adverse events | 16 weeks
  Safety will be assessed throughout the study by monitoring adverse events clinically and by Ultrasound imaging.

IPD SHARING:
Plan to Share IPD: No